CLINICAL TRIAL: NCT06675383
Title: SCREENING AFTER STROKE - ATRIAL FIBRILLATION - the SIGNIFICANCE of TIMING and CHOICE of DEVICE
Brief Title: SCREENING AFTER STROKE - ATRIAL FIBRILLATION
Acronym: SAS-AF
Status: Recruiting | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SAS-AF study
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial fibrillation screening in acute stroke
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples to a study-specific biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute ischemic stroke: Admitted with acute ischemic stroke and absence of atrial fibrillation on admission.

SUMMARY:
As much as 20-30% of all strokes are attributed to atrial fibrillation (AF), making the detection of AF highly important, as AF-related strokes are largely preventable with optimal treatment. Therefore, most guidelines recommend screening patients for AF after a stroke, although the optimal timing and choice of monitoring device for screening remain undefined. Our aim is to investigate whether AF screening as early as possible after stroke symptom onset provides a higher detection rate compared to screening after discharge. Additionally, we aim to determine if a 3-lead ECG device provides a higher detection rate compared to a 1-lead patch recorder.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most common cardiac arrhythmias, affecting over 2% of all adults in the general population, with prevalence increasing with age and cardiovascular risk factors. AF is responsible for at least 20% of all stroke cases, and stroke may often be the first manifestation of AF. Compared to strokes of other etiologies, AF-related strokes are associated with larger infarctions, worse outcomes, and higher mortality. Detecting previously undiagnosed AF in stroke patients is crucial for optimal secondary prevention through oral anticoagulation therapy.

As a result, guidelines emphasize the importance of AF screening in stroke patients to prevent recurrent strokes. Since AF can be asymptomatic and occur only intermittently, diagnosis may be easily missed or delayed. Studies have shown that prolonged screening increases detection rates. According to current knowledge, international AF and stroke guidelines recommend prolonged cardiac monitoring of at least 24 hours to detect subclinical AF if no other cause of stroke is identified.

However, while guidance exists on screening duration, none of the guidelines provide specific recommendations regarding the choice of device or the timing of screening. The sensitivity of AF detection likely depends on the screening strategy, timing, device, and algorithm used, but this area has been only minimally studied. Evidence suggests that the highest yield for AF detection may be early after stroke symptom onset. Nevertheless, significant knowledge gaps remain, and current screening strategies are not fully satisfactory.

Efforts to improve AF detection are warranted. This project aims to explore:

i. Whether prolonged AF screening initiated upon hospital admission after acute stroke results in a higher detection rate compared to prolonged ambulatory screening after discharge ii. Whether a 3-lead continuous ECG device has a higher detection rate compared to a 1-lead continuous patch recorder iii. A comparison of continuous vs. intermittent ECG AF screening for detection

The design involves a prospective observational trial of an unselected cohort of patients admitted with acute stroke to Bærum Hospital. Eligible participants include all patients above 18 years old without known AF or those with previously diagnosed paroxysmal AF exhibiting sinus rhythm upon admission. Upon admission to the Stroke Unit, patients will as soon as possible undergo a 48-hour in-hospital continuous heart monitoring, followed by a second 48-hour continuous heart monitoring upon discharge (ambulatory).

In addition, an intermittent AF screening with hand held thumb ECG, will be performed 3 times a day for 30 seconds, and for 3 consecutive days during the hospital stay in a sample of the participants, and compared to detection rate with continues heart monitoring.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Ischemic stroke
* Without known AF or those with previously diagnosed paroxysmal AF exhibiting sinus rhythm upon admission

Exclusion Criteria:

* AF at hosptial admission
* Unable or unwilling to provide informed consent
* A life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The design involves a prospective observational trial of an unselected cohort of patients admitted with acute stroke to Bærum Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of timing: Atrial fibrillation detection rate | 48 to 96 hours
  Detection rate of AF during initial in-hospital screening compared to detection rate during the second screening period starting at hospital discharge (ambulatory)

SECONDARY OUTCOMES:
Impact of device: Atrial fibrilation detection rate in 1-lead vs. 3-lead ECG recorder | 48 hours
  Will a 3-lead ECG device provide a higher detection rate compared to a 1-lead patch recorder when both devices are used in parallel on the same person
Impact of Continuity: Atrial fibrillation detection rate in continuous vs. intermittent ECG monitoring | 72 hours
  Will 48-hour continuous ECG monitoring provide a higher AF detection rate compared to intermittent AF screening using a handheld thumb ECG performed three times daily for 30 seconds over three consecutive days during the hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Håkon Ihle-Hansen, MD PhD, Study Director — Vestre Viken HF
Locations (1):
- Vestre Viken Hospital trust, Baerum Hospital, Sogneprest Munthe-kaas Vei 100, Gjettum, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Kamel H, Lees KR, Lyden PD, Teal PA, Shuaib A, Ali M, Johnston SC; Virtual International Stroke Trials Archive Investigators. Delayed detection of atrial fibrillation after ischemic stroke. J Stroke Cerebrovasc Dis. 2009 Nov-Dec;18(6):453-7. doi: 10.1016/j.jstrokecerebrovasdis.2009.01.012. PMID 19900647
- [Background] Tu HT, Campbell BC, Christensen S, Desmond PM, De Silva DA, Parsons MW, Churilov L, Lansberg MG, Mlynash M, Olivot JM, Straka M, Bammer R, Albers GW, Donnan GA, Davis SM; EPITHET-DEFUSE Investigators. Worse stroke outcome in atrial fibrillation is explained by more severe hypoperfusion, infarct growth, and hemorrhagic transformation. Int J Stroke. 2015 Jun;10(4):534-40. doi: 10.1111/ijs.12007. Epub 2013 Mar 12. PMID 23489996
- [Background] Sandercock P, Bamford J, Dennis M, Burn J, Slattery J, Jones L, Boonyakarnkul S, Warlow C. Atrial fibrillation and stroke: prevalence in different types of stroke and influence on early and long term prognosis (Oxfordshire community stroke project). BMJ. 1992 Dec 12;305(6867):1460-5. doi: 10.1136/bmj.305.6867.1460. PMID 1493391
- [Background] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Background] Kannel WB, Abbott RD, Savage DD, McNamara PM. Epidemiologic features of chronic atrial fibrillation: the Framingham study. N Engl J Med. 1982 Apr 29;306(17):1018-22. doi: 10.1056/NEJM198204293061703. PMID 7062992
- [Background] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399